CLINICAL TRIAL: NCT01952067
Title: Comparison of Two Cementing Techniques of the Femoral Component in a Hip Prosthesis. A Randomized Single-blind Trial
Brief Title: Comparison of Two Cementing Techniques of the Femoral Component in a Hip Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Kristiansund Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4.2008.1996
Record Dates: First submitted 2013-09-05; First posted 2013-09-27 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Hip
Keywords: Hip Prosthesis; surgery; cements; Radiostereometric Analysis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- line-to-line reaming (Experimental): Corail cemented femoral stem using line-to-line reaming and cementing technique, 28mm Alumine Biolox forte femoral head, Marathon cup
  Interventions: Procedure: line-to-line reaming and cementing technique
- standard over-reaming (Active Comparator): Corail cemented femoral stem using standard over-reaming with 2 broach sizes, 28mm Alumine Biolox forte femoral head, Marathon cup
  Interventions: Procedure: standard over-reaming with 2 broach sizes

INTERVENTIONS:
Procedure: line-to-line reaming and cementing technique
  Arms: line-to-line reaming
Procedure: standard over-reaming with 2 broach sizes
  Arms: standard over-reaming

SUMMARY:
The primary aim of the study is to compare migration of the cemented Corail stem representing polished surfaced versions of the femoral stem. Two different methods will be used for reaming the femoral canal and cementing of the stem. Radiostereometric analysis (RSA) will be used in migration measurements.

Furthermore pain, postoperative outcome and patient satisfaction will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring cemented primary total hip replacement.
* Patients with a diagnosis of osteoarthritis, avascular necrosis or post-traumatic arthritis
* Patients who understand the conditions of the study and are willing and able to comply with the post-operative scheduled clinical and radiographic evaluations and the prescribed rehabilitation
* Patient who signed the Ethics Committee approved specific Informed Consent Form prior to surgery

Exclusion Criteria:

* Patients who require revision of a previously implanted total hip replacement (THR)
* Patients who will receive a THR without cement
* Patients who have had a prior procedure of osteotomy on the femur
* Obese patients where obesity is severe enough to affect subject's ability to perform activities of daily living (body mass index, kg/m2: BMI >35)
* Patients with active or suspected infection
* Patients with malignancy

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Difference in subsidence of femoral stems of 200 microns | change from 6th day postoperative to 24 months
  Radiostereometric analysis (RSA) of implant migration: difference in translation and rotation (x-, y-, and z- axis) of the femoral stem

SECONDARY OUTCOMES:
Oxford Hip Score | change from 6th day postoperative to 24 months
  12 questions. Every question is scored 4 to 0 according to the selected response.
  Thus it is a continuous score ranging from 48-0. Each of the 12 questions on the Oxford hip score is scored in the same way with the score decreasing as the reported symptoms increase (ie. become worse). All questions are laid out similarly with response categories denoting least (or no) symptoms being to the left of the page (scoring 4) and those representing greatest severity lying on the right hand side (scoring 0).
EQ-5D-5L | change from 6th day postoperative to 24 months
  5 questions. Every question is scored 1 to 5 where 5 is worse outcome. For example one profile could be' 12233' We then convert this specific health state to an index value specific for that country. The index value calculator can be downloaded from the EuroQol Office. 5 questions. Every question is scored 1 to 5 where 5 is worse outcome. For example one profile could be' 12233' We then convert this specific health state to an index value specific for that country. The index value calculator can be downloaded from the EuroQol Office.
Harris Hip Score (HHS) | change from 6th day postoperative to 24 months
  Four subscales make up HHS. The first is pain, which measures pain severity (44 points); function, which is made up of daily activities and gait (47 points); the absence of deformity, which is a subscale that measures hip flexion, adduction, internal rotation, leg length discrepancy and range of motion measures.(4 points), and range of motion (5 points).
  The survey has 10 question items and scores range from 0-100 with higher scores representing less dysfunction and better outcomes.
Visual Assessment Scale (VAS) for pain | change from 6th day postoperative to 24 months
  A horizontal or vertical 10 cm line labelled at each end by descriptors such as 'no pain' and 'worse pain ever'. The patient marks the line to indicate pain severity and it is simply quantified by measuring the distance in cm from 0 (no pain) to the patient's marked rating.
Merle D'Aubigne scale | change from 6th day postoperative to 24 months
  The score includes the parameters pain, mobility, and ability to walk, with each rated from 0 points (worst condition) to 6 points (best condition). Addition of the scores for pain and mobility results in an absolute estimation of hip function.

CONTACTS AND LOCATIONS:
Overall Officials: Otto Schnell Husby, md phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- Kristiansund Hospital, Kristiansund, Norway

REFERENCES:
- [Result] Sevaldsen K, Schnell Husby O, Lian OB, Farran KM, Schnell Husby V. Is the French Paradox cementing philosophy superior to the standard cementing? A randomized controlled radiostereometric trial and comparative analysis. Bone Joint J. 2022 Jan;104-B(1):19-26. doi: 10.1302/0301-620X.104B1.BJJ-2021-0325.R2. PMID 34969272